CLINICAL TRIAL: NCT00174226
Title: Eight-Week, Double-Blind, 3-Arm Parallel, Placebo-Controlled, Randomized Efficacy And Safety Trial Of Atomoxetine, Atomoxetine Plus Buspirone, And Placebo In Adults With Attention Deficit Hyperactivity Disorder
Brief Title: Treatment of Adult ADHD With Atomoxetine or Atomoxetine and Buspar
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A9001245
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-07

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride; Buspirone

INTERVENTIONS:
Drug: Atomoxetine
Drug: Buspirone

SUMMARY:
Determine if there is a difference in treatment response for adults with ADHD who are treated with Strattera versus those treated with a combination of Strattera and buspirone

ELIGIBILITY:
Inclusion Criteria:

* Adults with ADHD

Exclusion Criteria:

* Other Axis I Psychiatric Disorders

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 241 (Actual)
Dates: Start 2004-11; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of Atomoxetine-Buspirone (ATX-BSP) vs placebo (PBO) and atomoxetine (ATX) monotherapy in adult patients with ADHD as measured by the mean change across 7 weeks in the Adult ADHD Investigator Symptom Rating Scale (AISRS) total score

SECONDARY OUTCOMES:
To characterize the safety over 8 weeks of ATX-BSP as compared to PBO and ATX monotherapy. To assess the response rate for the 3 treatment groups based on AISRS and CGI scores.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (8):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Woodstock, Vermont

REFERENCES:
- [Derived] Sutherland SM, Adler LA, Chen C, Smith MD, Feltner DE. An 8-week, randomized controlled trial of atomoxetine, atomoxetine plus buspirone, or placebo in adults with ADHD. J Clin Psychiatry. 2012 Apr;73(4):445-50. doi: 10.4088/JCP.10m06788. Epub 2012 Jan 10. PMID 22313788
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001245&StudyName=Treatment+of+Adult+ADHD+with+Atomoxetine+or+Atomoxetine+and+Buspar+